CLINICAL TRIAL: NCT03758547
Title: Physiological Effects of the Application of Secretion Removal Device in Invasively Ventilated Patients
Brief Title: Effects of Secretion Removal in Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Chief of Respiratory and Critical Care unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Stefano Nava
Record Dates: First submitted 2018-11-23; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Intervention Model Description: baseline (time0) application of 10 cycles of positive inspiratory and negative expiratory pressures (time1) application of percussion (time2)
Masking Description: patients deeply sedated and therefore not conscious
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- in-exufflator and percussion technique (Experimental): assess the physiological effects, of a "common" daily practice of secretion removal in intubated patients, that are: in-exufflator technique and percussion technique
  Interventions: Device: in-exufflator technique; Device: percussion technique

INTERVENTIONS:
Device: in-exufflator technique — application through a device of 10 cycles using positive pressure (30 cmH20) during inspiration and negative pressure (-30 cmH20) during exhalation
Device: percussion technique — sliding venturi system (phasitron), powered by compressed gas that can be changed from 0.8 up to 3.5 bar and that generates the oscillations in the range of 80-650 cycles/min

SUMMARY:
In this study the investigators will assess the effects of secretion removal on "noninvasive" respiratory mechanics, in deeply sedated mechanically ventilated patients All the mechanically ventilated patients will be submitted to the recording of compliance and resistance at baseline (time0), immediately after the application of 10 cycles alternating 30 cmH20 during expiration and -30 cmH20 during exhalation (time1). Afterward the patients will undergo an additional trail using the so called "percussion" technique, to assess any synergic effect of this procedure (time2)

DETAILED DESCRIPTION:
In this observational study, the investigators will assess the effects of two secretion removal techniques on passive respiratory mechanics, in patients undergoing invasive mechanical ventilation.

Consecutive patients will undergo 3 sequential assessments at time0 (baseline), at time1 after the application of of 10 cycles alternating 30 cmH20 during expiration and -30 cmH20 during exhalation and finally after a 20 sec application of a "percussion technique".

Protocol:

The patients will be ventilated without PEEP and sedated with a benzodiazepine infusion to produce complete relaxation and adaptation to the ventilator, as assessed by the complete absence of spontaneous efforts, so that there was no change in inspiratory flow rate, tidal volume, or respiratory rate during the three measurement periods.

Airway pressure (Paw) and flow (V) will be measured continuously throughout the respiratory cycle with the transducer and expiratory tidal volume will obtained by electrical integration of the flow signal.

Arterial blood gas specimens will be withdrawn from the radial artery and analyzed with a blood gas analyzer The patients will be studied in the semi recumbent position. After baseline measurements of respiratory mechanics will recorded under control conditions.

Direct measurement of PEEPi will be obtained using the following method:

After several breaths under controlled mechanical ventilation, and with the patient relaxed, the airway opening is occluded at the end of a tidal expiration, using the end-expiratory hold button incorporated in the ventilator.

The occlusion will be then released for the mechanical lung inflation, and after a few breaths the airway opening will be again occluded at the end of the inflation, using the end-inspiratory hold button of the ventilator.

The static compliance of the total respiratory system (Cst rs) will be corrected for the compliance of the ventilator tubing and the gas compression (0.8 ml/cm H20 2).

The end-inspiratory occlusion technique also allows determination of the inspiratory resistive properties of the respiratory system, named R,rs min and R,rsmax, that means the minimal respiratory resistances (those due mainly to the airways) and maximal respiratory resistances (those mainly due to stress relaxation and Pendelluft)

ELIGIBILITY:
Inclusion Criteria:

consecutive ventilated and intubated patients

1. age> 18 yrs
2. Sign inform consent
3. clinical indication for secretion removal from the endotracheal tube

   -

   Exclusion Criteria:
   * tracheotomy
   * bullous emphysema
   * pneumothorax

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in passive respiratory mechanics | immediate
  RESPIRATORY MECHANICS is monitored using the end-expiratory and end inspiratory technique, obtained pressing the hold command on the ventilator

SECONDARY OUTCOMES:
changes in arterial blood gases | immediate
  changes in arterial partial oxygen tension and in arterial partial carbon dioxide tension obtained with a puncture of the radial artery

IPD SHARING:
Plan to Share IPD: No
not allow to release individual data of the patients